CLINICAL TRIAL: NCT04865952
Title: Effect of Hyaluronic Acid Application in Gene Expression and Cellular Behavior 24-hours After Injury
Brief Title: Early Healing of Oral Soft Tissues: a Clinical and Biomolecular Analysis. Part III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea Pilloni MD DDS MS, Chairman Section of Periodontics Director of Master Program in Periodontics, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 5315 Prot 0640/2020
Record Dates: First submitted 2021-04-25; First posted 2021-04-29 (Actual); Last update posted 2022-10-04 (Actual); Status verified 2022-10

CONDITIONS: Wound Heal; Wound Surgical; Oral Soft Tissue Conditions; Hyaluronic Acid
Keywords: early wound healing; gingival tissue; wound healing; hyaluronic acid; soft tissue injury
MeSH Terms: conditions — Surgical Wound; Soft Tissue Injuries | interventions — Biopsy

STUDY DESIGN:
Intervention Model Description: split-mouth design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA application (treatment group - HA) (Experimental): periodontal surgery + HA application + buccal attached gingival (G) biopsies 24 hr after surgical procedure
  Interventions: Procedure: periodontal surgery + 24 hr buccal attached gingiva (G) biopsy; Other: HA application
- NO HA application (non treatment group - NT) (Other): periodontal surgery + buccal attached gingival (G) biopsies 24 hr after surgical procedure
  Interventions: Procedure: periodontal surgery + 24 hr buccal attached gingiva (G) biopsy

INTERVENTIONS:
Procedure: periodontal surgery + 24 hr buccal attached gingiva (G) biopsy — Periodontal surgery will be performed and 24 hr after the surgical procedure a 2mm punch biopsy will be harvested at the level of the buccal attache gingiva (G).
Other: HA application — HA will be applied at the end of the surgical procedure, at the level of the vertical released incisions (VRIs) and over VRIs
  Arms: HA application (treatment group - HA)

SUMMARY:
The purpose of the present study is to evaluate the effect of Hyaluronic acid application in the gene expression profile and cellular behavior in the early wound healing process -24 hours after injury- of the oral soft tissues.

DETAILED DESCRIPTION:
Although it has been demonstrated the role of HA in many different biological process related with tissue repair and regeneration, specific mechanisms involved in the early wound healing process in the oral soft tissues remains unclear.

A recent in vitro study evaluated the effects of two HA formulations on human oral fibroblasts involved in soft tissue wound healing/regeneration. The authors demonstrated that the investigated HA formulations maintained the viability of oral fibroblasts and increased their proliferative and migratory abilities. Moreover, enhanced expression of genes encoding type III collagen and transforming growth factor-β3, characteristic of scarless wound healing. Interestingly, TGFB1 remains unchanged. Moreover, compared to untreated control cells, either HA preparation upregulated the expression levels of COL3A1 in both HPFs and HGFs at 24 hour, whereas no effect on COL1A1 mRNA levels was detected The HAs upregulated the expression of genes encoding pro-proliferative, pro-migratory, and pro-inflammatory factors, with only a moderate effect on the latter in gingival fibroblasts. However, in vitro experiments have certain limitations. HA would undergo degradation to lower MW molecules following hyaluronidase activity during the post-operative period and will thus exert additional or even opposing effects on the wound repair process.28

To highlight, is the fact that in the latest years, the translational medicine focuses in research concerning scar-free wound healing tissues repair mechanisms and regarding this, it has been proposed that HA plays an important role in the fast and scarless fetal wound healing seeing during the first and second trimester.

Therefore, the aim of the present pilot study will be to evaluate the effect of hyaluronic acid application on gene expression and cellular behavior in the early wound healing process of gingival tissues. The second aim of the present work will be to evaluate the effect of HA in the wound healing clinical response.

Our hypothesis is that HA modifies the expression of genes related with the early wound healing response and the behavior of the main cells involved in this biological process: fibroblasts; stimulating and accelerating their wound healing potential.

ELIGIBILITY:
Inclusion Criteria:

* patients that required periodontal surgery;
* patients age between 30-60 years;
* patients with full mouth plaque score and full mouth bleeding score < 15%;
* patients with a good general healthy status;
* patients without any medicaments or drug consumption that can affect the healing process;
* non-smoking patients.

Exclusion Criteria:

* patients in pregnancy;
* patients in lactation period;
* patients with consumption of antibiotics or anti-inflammatory drugs in the previous six months;
* patients with systemic diseases.

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2021-04-29 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-06 (Actual)

PRIMARY OUTCOMES:
Changes from baseline fold regulation wound healing related genes at 24 hours HA application | 24 hours after surgery (T24 hours)
  Total RNA from biopsies or cell cultures was extracted using TRIzol reagent Quantitative real-time PCR (qRT-PCR) cDNA was generated and cDNA obtained were used for amplification of wound healing related genes using the appropriate TaqMan gene expression assay kits.
Clinical evaluation of early wound healing | 24 hours after surgery (T24 hours)
  Assessed with a clinical index (EHS- Early wound healing score). This score assessed clinical signs of re-epithelialization (CSR), clinical signs of haemostasis (CSH), and clinical signs of inflammation (CSI). Since complete wound epithelialization was the main outcome, the CSR score was weighted to be 60% of the total final score. Accordingly, a score of 0, 3, or 6 points was possible for the assessment of CSR, whereas scores of 0, 1, or 2 points were possible for CSH and CSI. Higher values indicated better healing. Accordingly, the score for ideal early wound healing was 10.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Pilloni, MD,DDS,MS, Study Director — University of Roma La Sapienza
Locations (1):
- Department of Oral and Maxillofacial Sciences. Section of Periodontics.Sapienza, University of Rome, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eming SA, Martin P, Tomic-Canic M. Wound repair and regeneration: mechanisms, signaling, and translation. Sci Transl Med. 2014 Dec 3;6(265):265sr6. doi: 10.1126/scitranslmed.3009337. PMID 25473038
- [Background] Warburton G, Nares S, Angelov N, Brahim JS, Dionne RA, Wahl SM. Transcriptional events in a clinical model of oral mucosal tissue injury and repair. Wound Repair Regen. 2005 Jan-Feb;13(1):19-26. doi: 10.1111/j.1067-1927.2005.130104.x. PMID 15659033
- [Background] Iglesias-Bartolome R, Uchiyama A, Molinolo AA, Abusleme L, Brooks SR, Callejas-Valera JL, Edwards D, Doci C, Asselin-Labat ML, Onaitis MW, Moutsopoulos NM, Gutkind JS, Morasso MI. Transcriptional signature primes human oral mucosa for rapid wound healing. Sci Transl Med. 2018 Jul 25;10(451):eaap8798. doi: 10.1126/scitranslmed.aap8798. PMID 30045979
- [Background] Wang Y, Tatakis DN. Human gingiva transcriptome during wound healing. J Clin Periodontol. 2017 Apr;44(4):394-402. doi: 10.1111/jcpe.12669. Epub 2017 Feb 11. PMID 28005267
- [Background] Vescarelli E, Pilloni A, Dominici F, Pontecorvi P, Angeloni A, Polimeni A, Ceccarelli S, Marchese C. Autophagy activation is required for myofibroblast differentiation during healing of oral mucosa. J Clin Periodontol. 2017 Oct;44(10):1039-1050. doi: 10.1111/jcpe.12767. Epub 2017 Aug 25. PMID 28646601
- [Background] Marini L, Rojas MA, Sahrmann P, Aghazada R, Pilloni A. Early Wound Healing Score: a system to evaluate the early healing of periodontal soft tissue wounds. J Periodontal Implant Sci. 2018 Oct 24;48(5):274-283. doi: 10.5051/jpis.2018.48.5.274. eCollection 2018 Oct. PMID 30405935
- [Background] Rojas MA, Ceccarelli S, Gerini G, Vescarelli E, Marini L, Marchese C, Pilloni A. Gene expression profiles of oral soft tissue-derived fibroblast from healing wounds: correlation with clinical outcome, autophagy activation and fibrotic markers expression. J Clin Periodontol. 2021 May;48(5):705-720. doi: 10.1111/jcpe.13439. Epub 2021 Feb 17. PMID 33527447
- [Background] Bansal J, Kedige SD, Anand S. Hyaluronic acid: a promising mediator for periodontal regeneration. Indian J Dent Res. 2010 Oct-Dec;21(4):575-8. doi: 10.4103/0970-9290.74232. PMID 21187628
- [Background] West DC, Hampson IN, Arnold F, Kumar S. Angiogenesis induced by degradation products of hyaluronic acid. Science. 1985 Jun 14;228(4705):1324-6. doi: 10.1126/science.2408340.
- [Background] Pilloni A, Bernard GW. The effect of hyaluronan on mouse intramembranous osteogenesis in vitro. Cell Tissue Res. 1998 Nov;294(2):323-33. doi: 10.1007/s004410051182. PMID 9799448
- [Background] Fujioka-Kobayashi M, Muller HD, Mueller A, Lussi A, Sculean A, Schmidlin PR, Miron RJ. In vitro effects of hyaluronic acid on human periodontal ligament cells. BMC Oral Health. 2017 Jan 16;17(1):44. doi: 10.1186/s12903-017-0341-1. PMID 28093072
- [Background] Nyman E, Henricson J, Ghafouri B, Anderson CD, Kratz G. Hyaluronic Acid Accelerates Re-epithelialization and Alters Protein Expression in a Human Wound Model. Plast Reconstr Surg Glob Open. 2019 May 1;7(5):e2221. doi: 10.1097/GOX.0000000000002221. eCollection 2019 May. PMID 31333952
- [Background] Asparuhova MB, Kiryak D, Eliezer M, Mihov D, Sculean A. Activity of two hyaluronan preparations on primary human oral fibroblasts. J Periodontal Res. 2019 Feb;54(1):33-45. doi: 10.1111/jre.12602. Epub 2018 Sep 27. PMID 30264516